CLINICAL TRIAL: NCT04607525
Title: Efficacy of Dexmedetomidine Infusion Without Loading Dose on Hemodynamic Variables and Recovery Time During Craniotomy: A Randomized Double Blinded Controlled Study
Brief Title: Dexmedetomidine Infusion Effect on Hemodynamic Variables During Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R 115 / 2020
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Hemodynamic Instability; Supratentorial Neoplasms
Keywords: Postoperative analgesia; Craniotomy; Dexmedetomidine
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D (Experimental): Group D: Patients received 0.5 µg/kg/h of Dexmedetomidine. Dexmedetomidine dosage was diluted in 50 ml syringe of normal saline
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): Patients received equal volume and rate of normal saline as Group D.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — On the scheduled time of operation, the head nurse opened each envelope just before surgery, prepared the infusion solution and handled it to the anesthesiologist who was blinded to the solution. He was then determined for collecting perioperative data.
  Group D: Patients received 0.5 µg/kg/h of Dexmedetomidine. Dexmedetomidine dosage was diluted in 50 ml syringe of normal saline Group C: Patients received equal volume and rate of normal saline as Group D.
  This dosing regimen was in accordance with existing guidelines [5] [6] [7].
  Arms: Group D
Drug: normal saline — On the scheduled time of operation, the head nurse opened each envelope just before surgery, prepared the infusion solution and handled it to the anesthesiologist who was blinded to the solution. He was then determined for collecting perioperative data.
  Group C: Patients received equal volume and rate of normal saline as Group D.
  Arms: Group C

SUMMARY:
There is no clear consensus among neuroanesthesiologists regarding which anesthetic regimen is optimal for craniotomy. Propofol and short-acting opioids (such as remifentanil, fentanyl, or sufentanil) are commonly used. However, use of opioids is associated with increased risk of respiratory depression and postoperative nausea and vomiting. Dexmedetomidine is a highly selective α2-adrenoreceptor agonist that has been considered as a useful and safe adjunct to anesthesia for various surgical procedures

DETAILED DESCRIPTION:
The investigators designed this randomized, double-blind study to evaluate the effectiveness of administration of Dexmedetomidine infusion at a dose of 0.5 µg/kg/h without loading dose during elective supratentorial craniotomy under GA. The investigators will compare intraoperative hemodynamics in both groups, intraoperative analgesic consumption, intraoperative blood loss, postoperative sedation scores, intraoperative need for rescue hypotensive agents, and finally the satisfaction of surgeons.

To our knowledge, the present study is the first to evaluate the effect of Dexmedetomidine infusion without loading dose in elective supratentorial craniotomy

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists- Physical status (ASA-PS) I and II patients,
* aged 18 to 65 years
* 70-80 kg
* both sexes
* undergoing elective supratentorial craniotomy for tumor resection

Exclusion Criteria:

* Patients under 18 years of age
* pregnancy,
* emergency surgery
* patients with a Glasgow Coma Score (GCS) less than 15.
* Those who had respiratory or cardiac dysfunction, renal insufficiency, liver impairment, or bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Mean areterial blood pressure | 4 to 8 hours
  incidence of intraoperative hemodynamic stability
Heart rate | 4 to 8 hours
  incidence of intraoperative hemodynamic stability
Number of Participants needed rescue agents | 4 to 8 hours

SECONDARY OUTCOMES:
Recovery time in minutes | At the end of operation
  Recovery time in minutes (time interval between discontinuation of isoflurane and extubation).
Postoperative sedation level | 1st 2 hours postoperatively
  Assessment of postoperative sedation level using "University of Michigan Sedation Scale (UMSS)" The UMSS is a simple observational tool that assesses the level of alertness on a five-point scale ranging from 1 (wide awake) to 5 (unarousable with deep stimulation). Score: 1- 5

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the study till 1 year
Access Criteria: Via email request